CLINICAL TRIAL: NCT00357929
Title: Weaning From Mechanical Ventilation Using Permissive Hypercarbia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kane High, Associate Professor of Anesthesiology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23214
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Respiration, Artificial; Respiratory Distress Syndrome, Adult
Keywords: permissive hypercarbia; weaning from mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Distress Syndrome

INTERVENTIONS:
Procedure: Permissive hypercarbia

SUMMARY:
Some patients receiving mechanical ventilation have difficulty weaning off the ventilator because of physiological factors such as pre-existing lung disease, respiratory distress syndrome, and trauma among others. Allowing patients to become hypercarbic (increased blood bicarbonate level) may make it easier for these patients to be taken off the ventilator and resume breathing on their own.

DETAILED DESCRIPTION:
The primary objective of this research is to assess the utility of permissive hypercarbia (PH) in the weaning of patients with risk factors for difficult weaning from mechanical ventilation. This pilot study seeks to validate the concept that PH will significantly improve the ability of patients to be weaned from mechanical ventilation and change the approach that physicians take to ventilator weaning for many patients.

Null Hypothesis: Patients with PH will not be weaned from mechanical ventilation more rapidly than those not receiving PH.

Patients with significant lung disease fail weaning from mechanical ventilation either as a result of an inability to oxygenate the blood or to adequately remove carbon dioxide. This results in longer Intensive Care Unit stays and increased morbidity and mortality as these patients have prolonged periods of mechanical ventilation. This study will focus on patients who have failure to adequately remove carbon dioxide (ventilatory failure) and endeavors to evaluate a method for enhanced carbon dioxide elimination by altering the acid-base status of the patients utilizing permissive hypercarbia (PH). PH will be used specifically during weaning from mechanical ventilation to enhance carbon dioxide elimination during this period. PH has used by some intensivists for this purpose but has not been critically evaluated in a clinical study.

Mechanical ventilation using PH maintains an increased CO2 with either partial or complete metabolic compensation. Therefore, the blood pH is either normal or slightly reduced. In patients who are adequately sedated, the reduced pH is well tolerated without respiratory distress or air hunger. However, if PH is to be used in awake patients as proposed here, full metabolic compensation would be required to avoid air hunger while being weaned from ventilator support. The metabolic compensation is produced either as a result of a renal compensation or, more typically in the ICU setting, iatrogenically. Metabolic alkalosis can be produced through the administration of alkalinizing agents or as a result of gastric suctioning or from contraction alkalosis resulting from the use of diuretics.

PH enhances CO2 elimination by increasing the concentration of CO2 in the exhaled gas. The pulmonary capillary pCO2 is elevated and therefore so is the alveolar CO2 and the exhaled or end-tidal CO2. Thus more CO2 is exhaled in an equal volume of exhaled gas. This increased CO2 concentration reduces the minute ventilation required to exhale the CO2 produced by the patient. PH will decrease the minute ventilation requirement even in patients with an increased dead space and will facilitate weaning these patients from mechanical ventilation by the same mechanism as just described.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 yo) patients in the intensive care units at the Hershey Medical Center who are on mechanical ventilation
* and whose clinical course permits weaning from mechanical ventilation
* and are felt to have risk factors for difficult weaning. (Risk factors will include patients with rib fractures, pulmonary contusions, obesity (BMI >30), or history of COPD or other significant lung disease.)
* all patients will have failed (rapid shallow breathing index >105) a 30 minute spontaneous breathing test.

Exclusion Criteria:

* Overt signs of sepsis including: a temperature > 38.5F, white blood cell count > 14000, systolic blood pressure < 100 mmHg,
* intracranial hypertension (ICP > 18 or based upon clinical exam and/or history),
* or pulmonary hypertension (by history or PAsys > 40 mmHg).
* or history of recent(past 6 mos)MI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-08; Primary Completion 2007-06-14 (Actual); Study Completion 2007-06-14 (Actual)

PRIMARY OUTCOMES:
Time for weaning from positive pressure support mechanical ventilation

SECONDARY OUTCOMES:
Percentage of subjects/group successfully weaned within seven days of trial participation

CONTACTS AND LOCATIONS:
Overall Officials: Kane M High, MD, Principal Investigator — Penn State University, College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States